CLINICAL TRIAL: NCT00234871
Title: A Phase IV, Randomized, Open-Label, Active Controlled Study to Compare the Effects of Tarka® and Lotrel® on Albuminuria in Hypertensive, Type 2 Diabetic Subjects With Diabetic Nephropathy
Brief Title: Tarka® vs. Lotrel® in Hypertensive, Diabetic Subjects With Renal Disease (TANDEM)
Acronym: TANDEM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Peter Bacher, MD, PhD, Abbott
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M03-599
Record Dates: First submitted 2005-09-13; First posted 2005-10-10 (Estimated); Last update posted 2008-07-15 (Estimated); Status verified 2008-07

CONDITIONS: Hypertension; Diabetes; Proteinuria
Keywords: Hypertension; Diabetes; Proteinuria; Tarka; Lotrel
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Proteinuria | interventions — trandolapril; Verapamil; benazepril; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: trandolapril/verapamil
- 2 (Active Comparator)
  Interventions: Drug: Lotrel (amlodipine/benazepril)

INTERVENTIONS:
Drug: trandolapril/verapamil — 2/180 mg QD with forced titration after 4 weeks to 4/240 mg QD
  Other Names: ABT-TARKA; Tarka
  Arms: 1
Drug: Lotrel (amlodipine/benazepril) — 5/10 mg QD with forced titration after 4 weeks to 10/20 mg QD
  Arms: 2

SUMMARY:
The primary objective of this study is to determine if trandolapril/verapamil (Tarka®) is superior to amlodipine/benazepril (Lotrel®) in reduction of albuminuria in hypertensive subjects with Type 2 diabetes mellitus (DM) and diabetic nephropathy

ELIGIBILITY:
Inclusion Criteria:

* Diabetes
* Hypertension
* Albuminuria

Exclusion Criteria:

* Type 1 DM.
* Subject has severe hepatic dysfunction at Screening as determined by liver function tests:

  * Bilirubin > 2.0 mg/dL.
  * ALT and/or AST > 3 times the upper limit of normal.
  * Subject has poorly controlled diabetes, based on HbA1c > 10% at Screening.
* Subject has non-diabetic renal disease.
* Subject has a hypersensitivity to ACE inhibitor, CCB, torsemide or sulfonylureas.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2004-01; Primary Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Changes in urinary albumin:creatinine ratio | 36 weeks

SECONDARY OUTCOMES:
Changes in blood pressure (BP), BP control, ABPM, proteinuria, GFR lipid parameters, glycemic control, quality of life, CRP, oxidative stress markers, clinical safety labs and adverse events. | 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Global Medical Information, Study Director — Abbott